CLINICAL TRIAL: NCT03402737
Title: Combined Hypofractionated Stereotactic Body Radiotherapy With Immunomodulating Systemic Therapy for Inoperable Recurrent Head and Neck Cancer: Detection of the Maximum Tolerated Dose.
Brief Title: SBRT + Immunomodulating Systemic Therapy for Inoperable, Recurrent H&N
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recrual.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Radiotherapie, Principal Investigator, University Hospital, Ghent
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/0636; 2017-000133-31 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2018-01-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Neoplasm
Keywords: Stereotactic body radiotherapy; Immunomodulating systemic therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: The range of dose-painting will be escalated in following levels:
  * 2x 6-8Gy
  * 3x 6-8Gy
  The standard "3+3" design will be used for the this trial. To obtain more precise toxicity rate of the MTD we will double the number of patients at the first dose prescription that gives totally 6 patients. The 3 remaining dose levels will include 3 patients each. Thus, fifteen (6+3+3+3) patients will be included in this radiotherapy dose finding study investigating the MTD.
  The number of patients will be doubled in case of 2 DLTs at the dose prescription I and 1 DLT at dose prescriptions II-IV with DLT in a maximum of 10 out of 30 patients.
  * 3x 6-10Gy
  * 3x 6-12Gy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic body radiotherapy + IM (Experimental): Single arm phase I trial with 3 Stereotactic Body Radiation Therapy dose-escalation arms.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — The range of dose-painting will be escalated in following levels:
  * 2x 6-8Gy (day 1-4)
  * 3x 6-8Gy (day 1-4-7)
  * 3x 6-10Gy (day 1-4-7)
  * 3x 6-12Gy (day 1-4-7)
  Patients will take cyclophosphamide orally 50 mg tablets, 1 tablet a day from the first day of irradiation for 8 consecutive weeks.
  Nivolumab will be considered as standard therapy in patients with cisplatin refractory locoregional disease recurrence. Nivolumab will be administered as per current standard of care. In case patients that are treated with nivolumab will be included in the trial, they will not be treated with cyclophosphamide.

SUMMARY:
To derive the maximum tolerated dose of hypofractionated stereotactic body radiotherapy (SBRT) using dose painting by numbers with immunomodulating systemic therapy in patients that are reirradiated for recurrent squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
The standard treatment in inoperable locally or regionally recurrent head and neck cancer has long been palliative systemic therapy using the so-called EXTREME-scheme: a combination of cisplatin, 5-fluorouracil and cetuximab. This therapy remains without realistic chances of cure. More recently, immunotherapy using nivolumab has demonstrated to result in long-term disease control of 1-2 year in cisplatin-refractory recurrent or metastatic head and neck cancer, however only in a small portion of patients (13%).

Fractionated high-dose local or regional re-irradiation is mostly given in a 6-7 weeks scheme. Using stereotactic body radiotherapy (SBRT), high radiotherapy doses can be given in a short time span. Severe late adverse events have been reported using SBRT but seem less frequent than in patients re-treated with conventional schedules. A possible solution to be able to administer higher doses is combining SBRT with dose painting, thus giving these high doses on small subvolumes only.

Addition of concomitant therapy to reirradiation may further improve outcomes due to radiosensitization and direct cytotoxicity. Therefore the investigator aims to combine high doses with concomitant therapy in the proposed study.

The immunomodulatory effect caused by radiation has been demonstrated both in animal models and clinical trials and leads to an enhanced local control as well as to eradication of distant metastasis. This so-called abscopal effect is reached through a systemic immune response evoked by the release of damage-associated molecular patterns (DAMPs) by the dying tumor-cells, also called immunogenic cell death (ICD).

The investigator hypothesizes that an abscopal effect could be present for patients presenting locoregional recurrent disease with asymptomatic distant metastases, thereby offering at least symptom control at the primary site while palliative systemic treatment could be postponed.

The proposed protocol focuses on patients with bad prognosis, as determined by a short timespan between primary therapy and recurrence (defined as 6-24 months after the end of the primary radiotherapy). It would bring the practical advantage of only 2-3 patient visits for the radiotherapy instead of ± 30-35 visits over 6-7 weeks. This shorter treatment schedule is expected to result in a direct gain in quality-of-life due to locoregional symptom control. It can also be expected that rescue systemic therapy will be postponed to a later stage of disease development, thereby prolonging overall survival.

The combination with systemic agents that are involved in immunogenic cell death bear the potential to result in a higher number of patients with longer periods of disease control and survival. The current standard of care, i.e. the combined systemic treatment with cisplatin - 5-fluorouracil - cetuximab, or nivolumab in case of former cisplatin use, can be used as a rescue regimen in case of therapy failure. In that sense, better overall survival from time of diagnosis of the index locoregional recurrent disease is expected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed local, regional or combined locoregional recurrence of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx or cancer of unknown primary (CUP) in the neck in previously irradiated tissue, with former irradiation with curative intent.
* Patients with non-symptomatic distant metastases and local, regional or combined locoregional recurrence can be included.
* In case of non-metastatic disease, the recurrence must be primarily unresectable recurrence and/or patients refused surgery.
* Time interval 6-24 months after the end of the initial radio(chemo)therapy for primary head and neck cancer.
* Decision of the Head and Neck Tumor Boards at the recruiting centre to offer salvage radio(chemo)therapy, palliative chemotherapy or anti-PD-1 antibody treatment with nivolumab for cisplatin-refractory locoregional recurrent head and neck squamous cell carcinoma.
* Karnofsky performance status ≥ 70.
* Age ≥ 18 years old.
* Informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* Previous radiotherapy was for cT1-2 cN0 M0 glottic cancer.
* Grade ≥ 4 late toxicity after the initial radio(chemo)therapy.
* Brachytherapy as treatment for second primary / recurrence.
* Previous (combination with) immunotherapy for the primary or the recurrent squamous cell carcinoma.
* Impossibility of oral intake of cyclophosphamide.
* For patients receiving cyclophosphamide: necessary intake during therapy of allopurinol, amiodarone, digoxin, hydrochlorothiazide, indomethacin, phenobarbital, phenytoin, warfarin. clopidogrel, ticlopidine, carbamazepine, efavirenz, rifampicin, ritonavir
* High risk for arterial blow-out: 1 of following criteria is sufficient to exclude patients:

  1. soft tissue necrosis
  2. skin invasion of the recurrent cancer
  3. circumferential involvement of > 180° of a carotid artery
* Symptomatic distant metastases.
* Other uncontrolled second primary tumors.
* Pregnant or lactating women.
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 3 months after radiotherapy
  maximum tolerated dose of hypofractionated stereotactic body radiotherapy (SBRT) using dose painting by numbers with immunomodulating systemic therapy in patients that are reirradiated for recurrent squamous cell carcinoma of the head and neck

SECONDARY OUTCOMES:
symptom palliation - pain | through study completion, an average of 12 months
  reduction in pain
symptom palliation - dysphagia | through study completion, an average of 12 months
  reduction in grade of dysphagia
local control | 3 months after SBRT and thereafter through study completion, an average of 12 months
  Assessment of:
  1. diameter of target lesion of SBRT (and, if present, non-target lesions) in mm
  2. tumor response according to recist criteria
Overall survival | through study completion, an average of 12 months
  To estimate overall survival
Progression free survival | through study completion, an average of 12 months
  To estimate progression-free survival
grade ≥ 3 toxicity-free survival | through study completion, an average of 12 months
  To estimate grade ≥ 3 toxicity-free survival (anemia, febrile neutropenia, fatigue, dysphagia, oral mucositis, laryngeal mucositis, pharyngeal mucositis, pharyngeal hemorrhage, pharyngeal necrosis, pharyngeal stenosis, pharyngolaryngeal pain, dry mouth)
QOL - general | before therapy, week 3, week 6, week 10, week 14
  To assess quality-of-life: EORTC QLQ
QOL - H&N specific | before therapy, week 3, week 6, week 10, week 14
  To assess quality-of-life: H&N35
topographic distribution of recurrence | through study completion, an average of 12 months
  To assess the topographic distribution of recurrence (inside/outside FDG-avid GTV)
time to further treatment | through study completion, an average of 12 months
  To assess time to further treatment
immune response | using serum taken before treatment and at each fraction of SBRT, at weeks 6-14
  To assess the immune response

CONTACTS AND LOCATIONS:
Overall Officials: Fréderic Duprez, MD, PhD, Principal Investigator — Gent University
Locations (3):
- Belgium (3):
  - Radiotherapy department, University Hospital Ghent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven
  - CHU Namur, Namur